CLINICAL TRIAL: NCT02055716
Title: A Randomised, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerance, Pharmacokinetics and Pharmacodynamics of Sulforadex® in Healthy Male Subjects Following Daily Dosing for 7 Days
Brief Title: Sulforadex in Healthy Human Males MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Evgen Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVG002N
Record Dates: First submitted 2014-01-29; First posted 2014-02-05 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- alpha-cyclodextrin (Placebo Comparator): A placebo comparator composed of the same acid resistant HPMC capsules filled with 300mg of alpha cyclodextrin
  Interventions: Drug: alpha-cyclodextrin
- Sulforadex (Experimental): 100mg or 300mg size 00 acid resistant HPMC capsules
  Interventions: Drug: Sulforadex

INTERVENTIONS:
Drug: Sulforadex
  Other Names: Stabilised sulforaphane
  Arms: Sulforadex
Drug: alpha-cyclodextrin
  Arms: alpha-cyclodextrin

SUMMARY:
To determine the safety and tolerability of multiple doses of Sulforadex® in healthy male volunteers over 7 days with qd or bid dosing

DETAILED DESCRIPTION:
This study will be conducted in a randomised, double-blind, placebo-controlled design with multiple ascending doses of Sulforadex® administered qd [once daily] or bid [twice daily]) to healthy male subjects between 18 to 45 years of age.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is a healthy male of any race aged 18 to 45 years, inclusive, at screening.
2. Subject has a BMI of 18 - 25 kg/m2 inclusive at screening.
3. Subjects must agree to use acceptable methods of contraception,
4. Subjects should not donate sperm from the time of the first administration of treatment or study medication until 3 months following administration of the last treatment or dose of study medication.
5. Subjects must be capable of understanding and complying with the requirements of the protocol and must have signed the ICF prior to undergoing any study-related procedures.

Exclusion Criteria:

1. All subjects must refrain from eating brassica vegetables or using brassica containing supplements for at least 7 days prior to the drug administration. Brassica vegetables include cabbage, cauliflower, horseradish, landcress, Ethiopian mustard, kale, collard greens, Chinese broccoli, brussels sprouts, Kohlrabi broccoli, broccoli flower, broccoli romanesco, wild broccoli, bok choy, Komatsuna, mizuna, rapini, flowering cabbage, Chinese cabbage, Napa cabbage, turnip root, rutabaga, canola/rape seed, Siberian kale, wrapped heart mustard cabbage, mustard seed (brown, black, white), tatsoi, rocket (arugula), garden cress, water cress, radish, daikon and wasabi.
2. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion.
3. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.
4. ECG abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis.
5. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, psychiatric, or other disease.
6. Positive results in any of the serology tests for Hepatitis B Surface Antigen (HbsAg), anti Hepatitis core antibody (anti HBc Ig G [and anti HBc IgM if IgG is positive], Hepatitis C virus antibodies (anti HCV), and human immunodeficiency virus HIV 1 and 2 antibodies (anti HIV 1/2).
7. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, tricyclic antidepressants and methadone) or from the alcohol breath test at screening and on admission (Day -1).
8. History or clinical evidence of alcohol or drug abuse.
9. Mentally handicapped.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 7 days
  Safety assessments will include standard laboratory safety tests (haematology, biochemistry, coagulation and urinalysis), vital signs, physical examinations, 12-lead ECG, telemetry and AE monitoring.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of sulforaphane | time 0, 30 min 1 2 4 8 12 & 24 hrs post dose on days 1,2 & 7
  Plasma sulforaphane concentrations will be measured by LCMS/MS assay.
  • Area under the plasma concentration-time curve from zero to time t of the last measured concentration above the limit of quantification (AUC0-t).

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Täubel, MD FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Limited, London, United Kingdom